CLINICAL TRIAL: NCT06376656
Title: Successful Ageing: Evidence-based Interventions to Delay Ageing-related Decline
Brief Title: Successful Aging and Age-related Decline
Acronym: MyAgeWell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunway University (Other)
Responsible Party: Principal Investigator, YookChin Chia, Professor, Head of Department of Medical Sciences, School of Medical and Life Sciences and Programme Leader of Postgraduate Diploma In Primary Care For Elderly, Sunway University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LRGS/1/2019/SYUC/02/1
Record Dates: First submitted 2024-04-03; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Aging; Elderly; Cognitive Decline; Physical Decline; Intervention Study
Keywords: Cognition; Physical Activity; Biological Aging; Intervention; Neuroscience; MRI; EEG; Biological Markers; Cost-benefit Analysis; Age-related Decline; Depression; Anxiety
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A cohort of older Malaysian adults will be recruited and assigned to one of the groups, either cognitive stimulation, physical activity, combined cognitive stimulation and physical activity, or non-intervention control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive stimulation (Experimental): Participants will take part in psychoeducation, videogaming, book club and technology training workshops.
  Interventions: Behavioral: Cognitive stimulation
- Physical activity (Experimental): Participants will take part in walking, Zumba, resistance exercise and aerobics sessions.
  Interventions: Behavioral: Physical activity
- Combined intervention (Experimental): Participants will take part in both cognitive stimulation and physical activity intervention sessions.
  Interventions: Behavioral: Cognitive stimulation; Behavioral: Physical activity
- Non-intervention control (No Intervention): Participants will not take part in any intervention.

INTERVENTIONS:
Behavioral: Cognitive stimulation — The cognitive stimulation will comprise of psychoeducation, videogaming, book club and technology training workshop sessions. Participants will take part in weekly sessions that are an hour long each.
  For every six months, the participants will alternate between psychoeducation, videogaming, book club and technology training workshop sessions.
  Arms: Cognitive stimulation; Combined intervention
Behavioral: Physical activity — The physical activity intervention will comprise of walking, Zumba, resistance exercise and aerobics sessions. Participants will take part in weekly sessions that are an hour long each.
  For every six months, the participants will alternate between walking, Zumba, resistance exercise and aerobics sessions until the end of intervention period.
  Arms: Combined intervention; Physical activity

SUMMARY:
Recent studies have shown promising cognitive and physical interventions aimed at slowing down ageing-related declines in quality of life, but they lack strong ecological validity (brief durations, unrealistic goals, no real-world application) and has yet to show robust evidence that such interventions are stable and suitable in the long-term. The investigators aim to examine whether these interventions can, over four years, significantly slow down the normal rate of ageing-related decline.

DETAILED DESCRIPTION:
This is a longitudinal, controlled, cohort study. The overarching aim in this intervention study is three-fold: (1) to test hypotheses derived from ageing-related theories, (2) to provide robust measurable evidence both in the long-term and validate meaningful interventions, and (3) provide quantifiable cost-benefit ratio to suggested solutions. A cohort of Malaysian older adults will be recruited and assigned to one of the groups, either cognitive stimulation, physical activity, combined cognitive stimulation and physical activity, or non-intervention control.

ELIGIBILITY:
Malaysian older adults aged 60 and above who fulfil the following criteria will be recruited:

Inclusion Criteria:

* Healthy and this includes those seeking regular medical attention,
* Have some form of mobility (ability to walk short distances at least 3m),
* Able to communicate in at least one of the following languages: English, Malay, Mandarin, Tamil.

Exclusion Criteria:

* Older adults with a history of stroke,
* Diagnosis of neurodegenerative diseases (such as Alzheimer's disease or Parkinson's) or psychiatric disorders,
* Uncorrected auditory and/or visual impairments,
* Currently on psychiatric medications,
* Immobile,
* Require full-time caregiver assistance,
* With comprehension impediments from the assessment portion of this project,
* A Montreal Cognitive Assessment (MoCA) score of <13.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive scores | 4 years
  Changes in cognitive scores will be evaluated using Montreal Cognitive Assessment (MoCA). Possible scores range from 0-30. Higher scores indicate less cognitive impairment.
Changes in electroencephalogram (EEG) | 4 years
  Onset of neural responses to errors in the Go/No Go task will be evaluated using EEG.
Changes in structural magnetic resonance imaging (MRI) | 4 years
  Relationship between Wisconsin Card Sorting Test performance and grey matter volume will be evaluated using structural MRI.
Cost-benefit analysis of intervention | 4 years
  The economic benefits from the interventions will be evaluated and will cover three aspects: financial, productivity and health.
Changes in levels of human salivary lactoferrin | 4 years
  Changes in levels of human salivary lactoferrin (ng/mL) will be measured using salivary Enzyme-Linked Immunosorbent Assay (ELISA) kits. Low levels of lactoferrin can potentially indicate higher risk for cognitive impairment.
Changes in levels of human salivary C-reactive proteins | 4 years
  Changes in levels of human salivary C-reactive proteins (CRP, mg/L) will be measured using salivary Enzyme-Linked Immunosorbent Assay (ELISA) kits. High levels of CRP can indicate inflammation and its association with greater cognitive decline.
Changes in salivary telomere length | 4 years
  Changes in salivary telomere length (T/S ratio) will be measured using quantitative PCR. A higher T/S ratio indicates better preservation of telomere length hence better preservation of cognition.

SECONDARY OUTCOMES:
Changes in depression scores | 4 years
  Changes in depression scores will be measured using part of the Center for Epidemiologic Studies Depression Scale (CES-D). Possible scores range from 0-42. Higher scores indicating greater frequency of depressive experiences.
Changes in anxiety scores | 4 years
  Changes in anxiety scores will be measured using part of the Form Y of the State-Trait Anxiety Inventory (STAI). Possible scores range from 6-24. Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Yook Chin Chia Professor, Datin, Dr, MBBS, FRCP, Principal Investigator — Sunway University; Tin Tin Su, Study Chair — Monash University; Rozainee Khairudin, Study Chair — The National University of Malaysia; Nur Ain Shahrier, Study Chair — Sunway University; Audrey Wei Ling Lim, Study Chair — Sunway University
Locations (1):
- Sunway University, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
No. However, limited access to data could be shared upon reasonable request.

REFERENCES:
- [Background] Bogataj S, Mesaric KK, Pajek M, Petrusic T, Pajek J. Physical exercise and cognitive training interventions to improve cognition in hemodialysis patients: A systematic review. Front Public Health. 2022 Oct 14;10:1032076. doi: 10.3389/fpubh.2022.1032076. eCollection 2022. PMID 36311587
- [Background] Erickson KI, Leckie RL, Weinstein AM. Physical activity, fitness, and gray matter volume. Neurobiol Aging. 2014 Sep;35 Suppl 2:S20-8. doi: 10.1016/j.neurobiolaging.2014.03.034. Epub 2014 May 14. PMID 24952993
- [Background] Murman DL. The Impact of Age on Cognition. Semin Hear. 2015 Aug;36(3):111-21. doi: 10.1055/s-0035-1555115. PMID 27516712
- [Background] Ogawa T, Hirose Y, Honda-Ogawa M, Sugimoto M, Sasaki S, Kibi M, Kawabata S, Ikebe K, Maeda Y. Composition of salivary microbiota in elderly subjects. Sci Rep. 2018 Jan 11;8(1):414. doi: 10.1038/s41598-017-18677-0. PMID 29323208
- [Background] Wells PM, Sprockett DD, Bowyer RCE, Kurushima Y, Relman DA, Williams FMK, Steves CJ. Influential factors of saliva microbiota composition. Sci Rep. 2022 Nov 7;12(1):18894. doi: 10.1038/s41598-022-23266-x. PMID 36344584
- [Background] Yong MH, Lawrie L, Schaefer A, Phillips LH. The Effects of Adult Aging and Culture on Theory of Mind. J Gerontol B Psychol Sci Soc Sci. 2022 Feb 3;77(2):332-340. doi: 10.1093/geronb/gbab093. PMID 34036302